CLINICAL TRIAL: NCT05234736
Title: A Phase 2 Study to Evaluate the Pharmacokinetic Profile of CBL-514 Injection in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetic Profile of CBL-514 Injection in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Caliway Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBL-0203
Record Dates: First submitted 2021-12-23; First posted 2022-02-10 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Subcutaneous Fat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CBL-514 (Experimental): All 10 participants enrolled in the study will receive a single course of treatment with CBL-514 800 mg (unit dose: 2.0 mg/cm^2) on the abdomen (administered as multiple subcutaneous injections) on Day 1 only.
  Interventions: Drug: CBL-514

INTERVENTIONS:
Drug: CBL-514 — CBL-514 800 mg (unit dose: 2.0 mg/cm^2)

SUMMARY:
This Phase 2 study will be an open-label and single course study to assess the safety, tolerability, PK and metabolite profile of CBL-514.

DETAILED DESCRIPTION:
This is a Phase 2 study to evaluate the safety, tolerability, PK and metabolite profile of CBL-514 injection at the maximal use dosage.

This Phase 2 study has an open-label and single course design. A total of 10 adult participants, composed of 5 females and 5 males, will be enrolled in a single cohort. Each participant will receive a single course of treatment with CBL-514 800 mg on the abdomen (administered as multiple subcutaneous injections) on Day 1 only.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female aged 18 years to 64 years old (at Screening), inclusive.
2. Body mass index (BMI) >18.5 and < 35 kg/m2 and body weight ≥ 50 kg at Screening and Day 1.
3. Participant has sufficient subcutaneous fat thickness of at least 3.00 cm (30.0 mm) measured by caliper skinfold method around treatment area at Screening and Day 1.
4. Voluntarily signs the Informed Consent Form (ICF) and, in the opinion of the Investigator or delegate, is physically and mentally capable of participating in the study, and willing to adhere to study procedures, including food and drink restrictions.

Exclusion Criteria:

1. Women of childbearing potential (WOCBP) who are not willing to commit to an acceptable contraceptive regimen from the time of Screening and throughout study participation until 90 days after the last IP dose, or who are currently pregnant or lactating. Male participants who are not willing to commit to an acceptable contraceptive method. Female participants who are not WOCBP are not required to use contraception.
2. Participant diagnosed with coagulation disorders or is receiving anticoagulant/antiplatelet therapy or medications or dietary supplements, which impede coagulation or platelet aggregation.
3. Participant has hemoglobin A1c (HbA1c) ≥ 9%, delayed wound healing, or any diabetic risks which, in the opinion of Investigator, is inappropriate to participate in the study.
4. Participant has a clinically significant cardiovascular disease and clinically significant abnormal findings in electrocardiogram (ECG).
5. Participant with active or prior history of malignancies within 5 years before Screening or being worked-up for a possible malignancy. Except adequately treated basal cell carcinoma of skin and in situ squamous cell carcinoma of skin would be eligible as per Investigator's discretion.
6. Participant with a history of human immunodeficiency virus (HIV)-1, hepatitis B, or hepatitis C infections or participants with active HIV, hepatitis B, or hepatitis C infections at Screening:
7. Participants with positive COVID-19 antigen test at Screening and Day 1.
8. Participants with any hepatic medical condition that, in the opinion of the Investigator, would compromise the participant's ability to undergo study procedures and/or interfere with the assessment of the obtained data.
9. Participants with a history of trypanophobia, the extreme fear of medical procedures involving injections or needles, or who experience vasovagal syncope and faint or pass out at the sight of blood or a needle.
10. Participant has abnormal skin or local skin conditions at the treatment area, which in the opinion of Investigator, is inappropriate to participate in the study, including but not limited to any of the following:
11. Participant who has the following procedures:

    1. Previous surgery which caused scar tissues on the anticipated treatment area before Screening or during the study,
    2. Liposuction to the region to be treated before Screening or during the study,
    3. Esthetic procedure e.g., cryolipolysis, ultrasonic lipolysis, LLLT, lipolysis injection to the region to be treated within 12 months before Screening or during the study.
12. Participant is undergoing chronic systemic steroid or immunosuppressive therapy.
13. Requiring continual use of the following therapeutic agents during the study: terfenadine, buspirone, fexofenadine, any medication that is known to strongly inhibit or induce CYP enzymes, sensitive CYP substrates or drugs with narrow therapeutic index, in the opinion of the Investigator, may affect the evaluation of the study product or place the participant at undue risk.

    If a participant needs to use the above-mentioned therapeutic agents during the study for any reason, these therapeutic agents should not be used for at least 2 days prior to dosing and until 1 day post-dose.
14. Unable to receive local anesthesia (e.g., history of hypersensitivity to lidocaine).
15. Participants with known allergies or sensitivities to the IP or its components.
16. Participants with liver cirrhosis or with inadequate liver function at Screening defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), total bilirubin (TBIL), or gamma-glutamyl transferase (GGT) > 3.0 × upper limit of normal (ULN).
17. Participants with any renal impairment, defined as abnormal serum creatinine, and urea > 1.5 × ULN or estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73 m2. Participants who are currently on dialysis should be excluded.

    Participants with an eGFR ≥ 60 and < 90 mL/min/1.73 m2 at Screening should be evaluated by the Investigator to exclude pre-existing renal disease or associated dysfunction. If mild decrease in eGFR is assessed by the Investigator as not clinically significant or not related to dysfunction, the subjects may be eligible upon the Investigator's assessment.
18. Use of other investigational drug or device within 4 weeks prior to Screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Assess maximum analyte concentration of CBL-514 in plasma (Cmax) | 12 time points on Day1 and Day2
  To evaluate maximum analyte concentration of CBL-514 in plasma (Cmax) after single dose injection.
Assess time to Cmax of CBL-514 in plasma (tmax) | 12 time points on Day1 and Day2
  To evaluate time to Cmax of CBL-514 in plasma (tmax) after single dose injection.
Assess area under the concentration-time curve of CBL-514 in plasma (AUC) | 12 time points on Day1 and Day2
  To evaluate area under the concentration-time curve of CBL-514 in plasma (AUC) after single dose injection.
Assess elimination half-life of CBL-514 in plasma (t1/2) | 12 time points on Day1 and Day2
  To evaluate elimination half-life of CBL-514 in plasma (t1/2) after single dose injection.
Assess apparent total plasma clearance of CBL-514 in plasma (CL/F). | 12 time points on Day1 and Day2
  To evaluate apparent total plasma clearance of CBL-514 (CL/F) after single dose injection.
Assess apparent terminal volume of distribution of CBL-514 in plasma (Vz/F). | 12 time points on Day1 and Day2
  To evaluate apparent terminal volume of distribution of CBL-514 in plasma (Vz/F) after single dose injection.

SECONDARY OUTCOMES:
Metabolites of CBL-514 in plasma | 12 time points on Day1 and Day2
  Identify and assess the metabolites of CBL-514 in plasma for the first 3 females and the first 3 males enrolled following administration of CBL-514 into subcutaneous fat.
Number of participants with treatment-related adverse events (TEAEs) as assessed by CTCAE v5.0 | Up to 4 weeks after last treatment
  Number of participants experiencing TEAEs by severity and relationship to investigational product (IP)
Number of participants with clinically significant abnormalities in anthropometric parameters | On Screening Day and Day1
  Anthropometric parameters include body height, body weight, and abdominal subcutaneous fat thickness.
Number of participants with clinically significant abnormalities in physical examination | Up to 2 weeks after last treatment
  Physical examination includes assessments of the cardiovascular, respiratory, gastrointestinal, dermatological, and neurological systems.
Number of participants with clinically significant abnormalities in clinical laboratory values | Up to 2 weeks after last treatment
  Clinical laboratory tests include Biochemistry, Hematology, Coagulation, Urinalysis, Virology and Pregnancy status test.
Number of participants with clinically significant abnormalities in vital signs | Up to 2 weeks after last treatment
  Vital signs measurements include body temperature, pulse rate, blood pressure, and respiratory rate.
Number of participants with clinically significant abnormalities in Electrocardiogram (ECG) | Up to 2 weeks after last treatment
  ECG parameters include heart rate, RR interval, PR interval, QT interval, QTc interval, and QRS interval.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sheu, Study Director — Caliway Biopharmaceuticals Co., Ltd.
Locations (1):
- DermResearch Inc, Austin, Texas, United States